CLINICAL TRIAL: NCT01603940
Title: Comparison Between Losartan and Benazepril in Diabetic Hypertensive Patients With Blood Pressure Not Controlled by Amlodipine: Effects on Echocardiographic Parameters, Vascular Stiffness and Endothelial Function.
Brief Title: Comparison Between Losartan and Benazepril in Diabetic Hypertensive Patients Not Controlled by Amlodipine
Acronym: CONTROL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Responsible Party: Principal Investigator, Ronaldo Altenburg Odebrecht Curi Gismondi, Investigator. Medical Doctor. Master of Sciences., Hospital Universitario Pedro Ernesto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONTROL STUDY
Record Dates: First submitted 2012-05-20; First posted 2012-05-23 (Estimated); Results first posted 2015-11-11 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Hypertension; Diabetes Mellitus
Keywords: Hypertension; Diabetes Mellitus; Vascular stiffness; Endothelial function
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — benazepril; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Losartan (Active Comparator): This group will receive 100 mg of losartan per day. Amlodipine will be maintained.
  Interventions: Drug: Losartan
- Benazepril (Active Comparator): This group will receive 20 mg of benazepril per day. Amlodipine will be maintained.
  Interventions: Drug: Benazepril

INTERVENTIONS:
Drug: Benazepril — Patients in this group will receive 20 mg of benazepril per day, orally, during 12 weeks.
  Other Names: Lotensin; 0078-0447-05
  Arms: Benazepril
Drug: Losartan — Patients in this group will receive 100 mg of losartan per day, orally, during 12 weeks.
  Other Names: Cozaar; 0006-0951-54
  Arms: Losartan

SUMMARY:
The purpose of this study is to compare losartan and benazepril in diabetic patients whose high blood pressure is not controlled by amlodipine and its relationship to statin current use.

DETAILED DESCRIPTION:
Hypertension and diabetes mellitus are important risk factors for cardiovascular morbidity and mortality. Endothelial dysfunction and vascular rigidity are two pathophysiological mechanisms that may explain this relationship. Recent publications showed that both ACEi (angiotensin-converting enzyme inhibitor-induced) and ARB (angiotensin receptor blocker) were capable of improving vascular stiffness and endothelial function, and that these effects occurred despite blood pressure reduction.

This study main objective is to assess if ARB (losartan) effects are different from ACEi (benazepril) in endothelial function in patients with diabetes mellitus type 2 and blood pressure not controlled by amlodipine and its relationship to statin current use.

Secondary analysis of vascular stiffness will be measured by pulse wave velocity and augmentation index. Echocardiographic parameters, such as indexes of diastolic function, will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatorial patients with age between 40 and 70 years-old.
* Systemic arterial hypertension previously diagnosed and in use of two or less anti-hypertensive drugs in the preceding 4 weeks.
* Type 2 diabetes mellitus in use of oral medication that were not changed in the preceding 4 weeks. Glycated hemoglobin A1c less than 9.0%.
* Accepted the consent form.

Exclusion Criteria:

* Office systolic blood pressure equal or more than 180 mmHg, with or without treatment
* Office diastolic blood pressure equal or more than 110 mmHg, with or without treatment
* Evidences of a secondary cause for hypertension
* Glycated hemoglobin A1c > 9.0%
* Insulin therapy
* Chronic kidney disease stage 4 or 5 or in dialysis
* Advanced target organ lesion, obtained by history or additional exams, and defined by: previous myocardial infarction, heart failure with ejection fraction less than 40%, cerebral vascular accident (ischemic or hemorrhagic), peripheral vascular disease (claudication or doppler with obstruction > 50% of vascular lumen), retinopathy with visual loss, symptomatic neuropathy.
* Cardiac arrhythmias, except for ectopic beats
* Any clinical or disabling condition that, in the opinion of the investigators, may confound or prejudice study results.
* Severe mitral regurgitation.
* Women in fertile age without contraceptive methods in use.
* Breastfeeding women.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wille Oigman, MD, DSc., Study Chair — Hospital Universitario Pedro Ernesto; Mario F Neves, MD, DSc., Study Director — Hospital Universitario Pedro Ernesto; Ronaldo A Gismondi, MD, MSc., Principal Investigator — Hospital Universitario Pedro Ernesto
Locations (1):
- Hospital Universitario Pedro Ernesto, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Gismondi RA, Bedirian R, Pozzobon CR, Ladeira MC, Oigman W, Neves MF. Renin-Angiotensin System Blockade Associated with Statin Improves Endothelial Function in Diabetics. Arq Bras Cardiol. 2015 Dec;105(6):597-605. doi: 10.5935/abc.20150123. Epub 2015 Oct 2. PMID 26465872

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Losartan | Benazepril
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan | Benazepril | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [53 to 63] | 57 [52 to 62] | 57 [52 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  Brazil | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Function
Description: Access endothelial function by brachial flow-mediated vasodilation (FMD) and compare it between groups (losartan and benazepril) and its relationship to current statin use.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of maximal vasodilation
Arm/Group | Losartan | Benazepril
Number analyzed (Participants) | 16 | 14
percentage of maximal vasodilation | 9.4 [7.7 to 13.5] | 8.8 [6.9 to 11.0]
Statistical Analysis 1: Comparison: Losartan vs Benazepril; Test type: Superiority or Other; p = 0.616, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Vascular Stiffness
Description: Access vascular stiffness by pulse wave velocity and compare it between groups (losartan and benazepril).
Time Frame: 12 weeks.
Measure: Median (Inter-Quartile Range); unit: m/s
Arm/Group | Losartan | Benazepril
Number analyzed (Participants) | 16 | 14
m/s | 8.5 [7 to 9.7] | 8.5 [7.8 to 9.4]
Statistical Analysis 1: Comparison: Losartan vs Benazepril; Test type: Superiority or Other; p = 0.28, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Systolic Blood Pressure
Description: Compare both groups effects on systolic blood pressure.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Losartan | Benazepril
Number analyzed (Participants) | 16 | 14
mmHg | 134 [127 to 143] | 139 [130 to 154]
Statistical Analysis 1: Comparison: Losartan vs Benazepril; Test type: Superiority or Other; p = 0.618, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Diastolic Blood Pressure
Description: Compare both group effects on diastolic blood pressure.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Losartan | Benazepril
Number analyzed (Participants) | 16 | 14
mmHg | 80 [69 to 84] | 82 [74 to 89]

5. Secondary Outcome: Vascular Stiffness by Augmentation Index
Description: Estimate vascular stiffness by measuring augmentation index and compare it between losartan and benazepril groups.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of augmentation pressure
Arm/Group | Losartan | Benazepril
Number analyzed (Participants) | 16 | 14
percentage of augmentation pressure | 28 [21 to 37] | 35 [26 to 41]

ADVERSE EVENTS:
Arm/Group | Losartan | Benazepril
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 2/16 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=16) | Benazepril (N=14)
Edema (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Not severe edema in losartan group.
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cough due to benazepril (ACEi: angiotensin-converting enzyme inhibitor-induced)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No